CLINICAL TRIAL: NCT07219914
Title: Akashic Records and Mental Health Outcomes
Brief Title: This Study Explores the Mental Health Impact of Two Akashic Records Sessions.
Acronym: Akashic Record
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rasa Healing Inc (Other)
Responsible Party: Principal Investigator, Candice Rasa, LCSW, Akashic Records Facilitator, Therapist, Rasa Healing Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: #2024-0199
Record Dates: First submitted 2025-10-18; First posted 2025-10-22 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Resilience; Connectedness; Depression; Anxiety; Stress
Keywords: mental health; anixety; depression; stress; resilience; connectedness; transpersonal psychology; spirituality; past lives; akashic records; akashic field; exploratory pilot study; altered states
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Single-arm pilot study: all participants receive two Akashic Records sessions (one 90-minute and one 50-minute) and complete validated clinical scales at baseline, post-session, and 60-day follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Akashic Records Session Arm (Experimental): All participants receive two Akashic Records sessions: one 90-minute session and one 50-minute session, delivered virtually by a licensed clinician. Participants also complete validated clinical scales at baseline, post-session, and 60-day follow-up.
  Interventions: Behavioral: Akashic Records Session

INTERVENTIONS:
Behavioral: Akashic Records Session — Participants will receive two individual Akashic Records sessions. The first session lasts 90 minutes and the second session lasts 50 minutes. Sessions are conducted virtually by a licensed clinician trained in Akashic channeling. Participants are encouraged to set intentions, receive channeled information, and reflect on insights
  Other Names: Akashic Channeling; Akashic Reading; Akashic Field Channeling

SUMMARY:
The goal of this clinical study is to learn the impact of two Akashic Records sessions on mental health symptoms in adults. We want to see how sessions are linked to stress, anxiety, and depression, and to resilience (ability to bounce back) and feelings of connectedness (to self, community, and humanity).

Main questions this study will answer are:

After two sessions, what is the impact on stress, anxiety, and depression? After two sessions, what is the impact on resilience and connectedness? How do participants describe their experience of the sessions? After two sessions, what are participants' views of their problems (insight), emotional experiences (impact) and observable behaviors in their daily life?

What participants will do:

Complete online surveys about their mood at four points: before the first session, before the second session, after the second session, and again 2 months later.

Surveys include:

DASS-21 (Depression, Anxiety, and Stress Scale) CD-RISC-10 (Connor-Davidson Resilience Scale) WATTS (Connectedness Scale) A short demographic form and satisfaction survey

Attend two individual Akashic Records sessions (50-90 minutes each) over private video platform with a licensed clinical social worker (principal investigator) The first 50 participants will also join a one-hour interview with open ended questions with a licensed clinical social worker (co-investigator) about one week after the second session to share their experience in their own words.

Who can take part:

Adults ages 18 and older who can read and consent in English and who have experienced stress, anxiety, or low mood in the past year.

How the research will happen:

Sessions are held by secure video call. Participants will also complete private online surveys before, during, and after the sessions. Some participants may be invited to share their experiences in a one-on-one interview. All information is kept private and names are removed before analysis.

Risks and benefits:

Talking about personal topics may bring up strong emotions. Licensed clinicians conduct sessions, offer support, and provide referrals if needed.

Possible benefits include new insights, greater peace or meaning, and improved coping; benefits are not guaranteed.

Why this matters:

Many people seek spiritual or transpersonal support for emotional concerns. This pilot study will provide early evidence on whether Akashic Records sessions may be a helpful, low-risk option and will guide future research.

DETAILED DESCRIPTION:
The study aims to address the following research question: How do Akashic Records sessions impact mental health as evidenced by changes in self-reported stress, anxiety, and depression, and changes in resilience and connectedness?

This study is a single-arm, mixed-methods, exploratory pilot trial designed to evaluate the effects of Akashic Records sessions on mental health outcomes. The intervention consists of two individual sessions (one 90 minutes and one 50 minutes) delivered virtually by a licensed clinical social worker trained in Akashic Records channeling.

All participants are assigned to the same intervention arm consisting of two Akashic Records sessions; the study does not include randomization or a control/comparator group. To reduce potential confounding, participants are instructed to notify the research team of any changes in their mental health care or spiritual practices during the study period. They are also asked to maintain stability in their usual activities within these domains to support interpretability of pre-post outcomes.

The sessions follow a standardized structure to ensure reproducibility. Each session begins with an opening procedure that includes a brief Akashic prayer and a short reflection period for intention-setting. During the channeling process, the clinician conveys impressions received through intuitive modalities such as imagery (clairvoyance), auditory impressions (clairaudience), empathic resonance (clairsentience), and cognitive impressions (claircognizance). Information is verbalized in real time, and participants are invited to reflect, ask questions, and engage in dialogue to deepen integration. The clinician provides empathic support and reflective listening but does not apply structured psychotherapeutic interventions. Sessions conclude with a structured summary, identification of participant takeaways, and a formal closing statement.

The primary focus is on changes in validated clinical scales: the Depression, Anxiety, and Stress Scale (DASS-21), the Connor-Davidson Resilience Scale (CD-RISC-10), and the WATTS Connectedness Scale. Assessments are collected at four timepoints: baseline (T0), prior to the second session (T1), after the second session (T2), and 60 days following the intervention (T3).

In addition to quantitative endpoints, qualitative data are obtained from semi-structured interviews conducted with the first 50 participants until data saturation is reached. These interviews explore participant motivations, perceived benefits, integration of insights, and challenges. Transcripts are analyzed using structural and in vivo coding, followed by thematic analysis to generate emergent themes.

Approximately 100 adults will be enrolled, with inclusion criteria requiring age 18 or older, ability to provide informed consent, and willingness to engage in discussion of personal and emotional themes. Exclusion criteria include substance use disorder within the past 12 months, psychotic disorders, active suicidal ideation, or prior Akashic Records sessions within the past six months.

This research is conducted under expedited review and approval by Pearl IRB. Data are collected via HIPAA-compliant platforms (Jotform, Google Meet, and Dedoose), de-identified with unique participant IDs, and securely stored in encrypted systems.

The principal investigator will deliver all Akashic Records sessions but will not have access to raw survey data, qualitative transcripts, or primary statistical outputs, thereby reducing potential bias. The co-investigator will conduct prescreen interviews, review informed consent with participants, administer semi-structured interviews, and lead the qualitative analysis process with support from the independent research team. The research coordinator will manage participant communications, distribute validated clinical scales at designated timepoints, monitor adherence to study timelines, and ensure data is securely collected and logged.

This study is the first formal attempt to evaluate the Akashic Records in a structured clinical research design. Findings are intended to provide foundational evidence and inform the design of future controlled studies examining transpersonal and nonlocal interventions as potential contributors to mental health outcomes.

ELIGIBILITY:
Inclusion:

* 18 years old and over
* Ability and willingness to provide written, informed consent in English prior to initiation of any study-related procedures and adhere to all study requirements
* Willingness to engage in discussion about past life patterns and emotions
* Self-report of anxiety, depressive or stress symptoms in the last 12 months

Exclusion:

* Inability to provide consent due to cognitive impairment, mental health disorders, or other conditions that impact their ability to understand the nature, risks, and benefits of the study.
* History of alcohol or substance use disorder within 12 months
* History of hypomania or psychotic episode within 12 months
* Prior history (lifetime diagnosis) of schizophrenia spectrum, or other psychotic disorders
* Experiencing any other serious mental or physical health issues that would impact their ability to engage in the research study
* Has either attempted suicide, has documented medical history of suicidal ideation, or been hospitalized due to suicide risk within 1 year prior to prescreening.
* Previous Akashic Record Session with Interventionist, Candice S. Rasa, LCSW or previous Akashic Record Session with any other provider within 6 months.
* Any form of medicinal therapy should be stable 3 months prior to screening with no plan to start, stop or alter the use of any prescribed medications, supplements or other therapies from informed consent
* Any form of non-medical therapy should be stable 3 months prior to pre-screening with no plan to start, stop or alter use of psychotherapy, acupuncture, hypnosis, or other similar therapy from the time of providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-11-22 (Estimated); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
DASS-21 (Depression, Anxiety, Stress) Clinical Scale | T0: Baseline and 7 days before 1st session (Session #1 is within 30 days of prescreen). T1: No more than 7 days before 2nd session (Session #2 is 10-21 days after 1st). T2: Within 7-14 days after 2nd session. T3: Within 60-80 days after 2nd session
  Change in participant self-reported depression, anxiety, and stress symptoms as measured by the DASS-21 (Depression, Anxiety, Stress Scale - 21 items). The DASS-21 has three subscales (Depression, Anxiety, Stress), each ranging from 0-42. Higher scores indicate greater symptom severity. Scores are calculated by summing responses (0 = "did not apply to me at all" to 3 = "applied very much/most of the time") and multiplying by two for comparability with the original 42-item scale. Analysis will compare baseline to post-intervention values across timepoints. The DASS-21 will be given to participants at 4 time points during the study.

SECONDARY OUTCOMES:
CD-RISC-10 (Resilience) Clinical Scale | T0: Baseline and 7 days before 1st session (Session #1 is within 30 days of prescreen). T1: No more than 7 days before 2nd session (Session #2 is 10-21 days after 1st). T2: Within 7-14 days after 2nd session. T3: Within 60-80 days after 2nd session
  Change in participant self-reported resilience as measured by the CD-RISC-10 (Connor-Davidson Resilience Scale - 10 items). Scores range from 0-40, with higher scores indicating greater resilience (ability to adapt and bounce back from stress). Each item is scored 0 ("not true at all") to 4 ("true nearly all the time"). Total scores are calculated by summing item responses. Analysis will compare baseline to post-intervention values across timepoints. The CD-RISC-10 will be given to participants at 4 time points during the study.
WATTS Connectedness Scale | T0: Baseline and 7 days before 1st session (Session #1 is within 30 days of prescreen). T1: No more than 7 days before 2nd session (Session #2 is 10-21 days after 1st). T2: Within 7-14 days after 2nd session. T3: Within 60-80 days after 2nd session
  Change in participant self-reported connectedness as measured by the WATTS Connectedness Scale. This validated scale assesses three domains of connectedness: to self, to others, and to the wider world/humanity. Items are rated on a 0-100 scale, with higher scores indicating stronger connectedness. Total and subscale scores are calculated as means of item responses. Analysis will compare baseline to post-intervention values across timepoints. The WATTS will be given to participants at 4 time points during the study.

OTHER OUTCOMES:
Participant Satisfaction Survey (Feasibility/Acceptability) | T2 (7-14 days after the second session, prior to the semi-structured interview)
  Participant satisfaction with the Akashic Records sessions, assessed using a 5-point Likert scale (1 = very dissatisfied to 5 = very satisfied). Higher scores indicate greater satisfaction and acceptability of the intervention. Results will be summarized descriptively (means, standard deviations, frequencies) to evaluate feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Candice S Rasa, LCSW, Principal Investigator — Rasa Healing Inc
Locations (1):
- Virtual/ No Physical Facility, Palm City, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No, individual participant data (IPD) will not be shared due to the sensitive nature of qualitative interviews and personal health information. Only de-identified, aggregated data will be accessible to research analysis personnel outside the core team (PI, Co-PI, and Research Coordinator). Published results and peer-reviewed articles will report only group-level findings and representative de-identified quotes, with no individual-level data disclosed.

REFERENCES:
- [Background] Sheldrake R. An experimental test of the hypothesis of formative causation. Riv Biol. 1992;85(3-4):431-43. PMID 1341836
- [Background] Laszlo, E. (2007). Science and the Akashic Field: An Integral Theory of Everything. Inner Traditions.
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Watts, R., et al. (2017). Patients' accounts of increased "connectedness" and "acceptance" after psilocybin for treatment-resistant depression. Journal of Humanistic Psychology, 57(5), 520-564. https://doi.org/10.1177/0022167817709585
- [Background] Rubik B, Muehsam D, Hammerschlag R, Jain S. Biofield Science and Healing: History, Terminology, and Concepts. Glob Adv Health Med. 2015 Nov;4(Suppl):8-14. doi: 10.7453/gahmj.2015.038.suppl. Epub 2015 Nov 1. PMID 26665037
- [Background] Brysbaert M. How Many Participants Do We Have to Include in Properly Powered Experiments? A Tutorial of Power Analysis with Reference Tables. J Cogn. 2019 Jul 19;2(1):16. doi: 10.5334/joc.72. PMID 31517234
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174

DOCUMENTS (3):
  • Study Protocol (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT07219914/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT07219914/SAP_001.pdf
  • Informed Consent Form (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT07219914/ICF_002.pdf